CLINICAL TRIAL: NCT02143076
Title: Use of WISE Device Technology to Measure Medication Adherence in Youth With Sickle Cell Disease (SCD): A Pilot Study
Brief Title: Medication Adherence in Youth With Sickle Cell Disease (SCD)
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WISEP
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Sickle Cell Disease
Keywords: Medication Adherence; Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sickle Cell Disease: Participants will complete three questionnaires during the course of the study: Demographic Questionnaire, Medical Adherence Measure Questionnaire, and Acceptability Questionnaire. All questionnaires will be completed in a private clinic room.
  Interventions: Behavioral: Demographic Questionnaire; Behavioral: Medical Adherence Measure Questionnaire; Behavioral: Acceptability Questionnaire

INTERVENTIONS:
Behavioral: Demographic Questionnaire — At study enrollment, participants will complete a questionnaire to collect demographic information about the participant's family background, education and living situation.
Behavioral: Medical Adherence Measure Questionnaire — At the two-month follow-up visit, participants will be asked to complete a questionnaire describing all medications prescribed for them, when they take their medications, how much medication they take each time, how many times during the week they missed taking or were late taking each medication, reasons why they missed or were late, and how they manage their medications.
  In the case that a participant's clinic schedule is delayed greater than two months from the time of consent (e.g., missed appointment, change in clinic appointment frequency), procedures scheduled for the anticipated 2-month visit will take place at the participant's next clinic appointment.
Behavioral: Acceptability Questionnaire — At the two-month follow-up visit, participants will be asked to complete a questionnaire about their perceptions of using the Wise electronic medication container.
  In the case that a participant's clinic schedule is delayed greater than two months from the time of consent (e.g., missed appointment, change in clinic appointment frequency), procedures scheduled for the anticipated 2-month visit will take place at the participant's next clinic appointment.

SUMMARY:
Youth diagnosed with sickle cell disease (SCD) may have difficulty taking medication as prescribed (adherence). Hydroxyurea (HU) is one medication that youth may take to help manage SCD. Electronic adherence monitoring is widely considered the gold standard in objective adherence measurement. These monitors provide continuous, real-time records of medication adherence and reveal problematic behavior patterns, including underdosing, overdosing, delayed dosing, "drug holidays" (i.e. where individuals do not take medications for a specified interval of time), and "white coat" adherence (i.e., a pattern of drug adherence as a function of time where individuals display good adherence immediately before and after clinic attendance with worsening adherence in the period between).

Overall, electronic adherence measures are considered valid, reliable, and accurate, with clear advantages over pharmacy refill records, physician estimates and self-report measures. Currently, only one electronic measure capable of monitoring medications in both pill and liquid form is being manufactured: WisePill and WiseBag. While data are limited regarding its validity and reliability, preliminary data support the use of Wise technology to measure adherence to medication. The current study will determine the Wise device's ability to feasibly measure adherence to liquid and solid form HU medication in a pediatric SCD population.

DETAILED DESCRIPTION:
This research study will evaluate HU adherence using an electronic storage device (Wise device) compared to caregiver report, youth report, lab values, and pill-count adherence measures. The investigators will ask participants to store their medication in the Wise device and answer questions about their use of the device during normal clinical care visits.

PRIMARY OBJECTIVE

* To examine feasibility of the WISE device by estimating a) rate of consent to the study, b) rate of WISE device use, c) rate of WISE device failure, and d) the perceived acceptability of using the WISE device, as reported by caregivers and youth.

SECONDARY OBJECTIVE

* To estimate the association between HU adherence as measured by the Wise device, to a) caregiver-report, b) youth-report, c) lab values, d) pill-count, and e) Medication Possession Ratio (MPR) adherence measures.

Evaluation of study outcomes will be stratified by age group: (1) infants/toddlers, ages 0-7 years; (2) school age, ages 8-12 years; and (3) teen, ages 13-17 years.

At study enrollment, participants will be asked to complete one questionnaire and will receive instructions on how to use the Wise device. They will be asked to use the Wise device over the following two months. A study team member will contact each participant by phone within seven days of study enrollment to monitor participant use of the Wise device and to answer any questions. Participants will be asked to return the Wise device in two months at their normal clinic care visit. At this visit, participants will be asked to complete two more questionnaires and, as part of standard clinical care, a pill count/bottle weight will be completed by the pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCD (any genotype).
* Less than 18 years of age at time of study entry.
* Currently followed in the St. Jude Children's Research Hospital (SJCRH) SCD clinic.
* Stable HU dose prescribed (in pill or liquid formulation) for ≥ 6 months without documented hematological toxicity (excluding dose adjustments for weight gain).
* Lives with their primary caregiver.
* Anticipated to return to clinic at proposed 4-week or 8-week intervals.

Exclusion Criteria:

* Primary caregiver and/or youth unable to understand English and/or youth not cognitively intact (known IQ < 70) such that the study questionnaire cannot be understood and completed.
* Any condition or chronic illness that in the opinion of the PI or Co-I makes participation on the study ill-advised.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will have a diagnosis of sickle cell disease,be receiving treatment with hydroxyurea, and meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percent Rate of Consent to Study Participation | Baseline
  Of the total number of eligible participants, the percent of participants who agree to participate.
Percent Rate of Device Use | Two months after baseline
  The percent of the total participants who keep medicine in the device during the entire trial period.
Percent Rate of Device Failure | Two months after baseline
  Percent of devices that failed defined as a device does not register opening as verified by study staff at the time device is returned to the study team.
Acceptability of Using the Wise Device | Two months after baseline
  Responses by participants and/or caregivers to the Acceptability Questionnaire based on the Likert scale from strongly disagree to strongly agree.

SECONDARY OUTCOMES:
Medication Adherence as Measured by Wise Device Compared to Other Measures of Medication Adherence | Two months after baseline
  Adherence will be determined and compared between: a) adherence indicated by Wise device, b) adherence indicated by caregiver and youth-report, c) adherence indicated by lab values, d) adherence indicated by pill count/bottle volume, and e) adherence indication by medication possession ratio (MPR).
  Each participant's Wise adherence will be calculated as: [(number of device openings ÷ medication prescribed) x 100] where larger percentages suggest better adherence (range: 0-100%). Descriptive statistics for Wise device adherence and other adherence measures, including mean and standard deviation, median and interquartile range, will be estimated. Spearman's rank correlation coefficients and intraclass correlations between different adherence measures will be calculated to measure the associations between HU adherence measures for the entire sample as well as for each age group.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ingerski, PhD, Principal Investigator — St. Jude Children's Research Hospital; Jerlym Porter, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols